CLINICAL TRIAL: NCT02172430
Title: A Multiple Dose Comparison of Tiotropium 18 μg Inhalation Capsules and Oxitropium MDI (2 Puffs of 100 μg) in a One-year, Open-Label, Safety and Efficacy Study in Patients With COPD
Brief Title: Comparison of Tiotropium Inhalation Capsules and Oxitropium Metered Dose Inhalator (MDI) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205.227
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Tiotropium (Experimental)
  Interventions: Drug: Tiotropium powder inhalation capsules
- Oxitropium bromide (Active Comparator)
  Interventions: Drug: Tersigan®

INTERVENTIONS:
Drug: Tiotropium powder inhalation capsules — Powder inhalation via the HandiHaler® once daily
  Arms: Tiotropium
Drug: Tersigan® — 2 puffs of oxitropium three times daily via MDI
  Arms: Oxitropium bromide

SUMMARY:
The objective of this study is to investigate the long-term safety of Ba 79 BR (tiotropium) powder inhalation in patients with COPD using oxitropium bromide (Tersigan) as a comparator. Secondarily, the long-term efficacy of Ba 679 BR is also investigated

ELIGIBILITY:
Inclusion Criteria:

The patients with COPD (chronic bronchitis, emphysema) whose symptoms are stable and who satisfy the following criteria

1. Patients with FEV1.0 of <=70% of predicted normal and FEV1.0/FVC of <=70% in the screening test (The FEV1.0 value should also be <=70% of predicted normal on the starting day of administration (visit 2).)
2. Patients with a smoking history (<number of cigarettes smoked a day x number of smoking years> is >=200.)
3. Male or female patients aged >=40 years old

Exclusion Criteria:

1. Patients complicated with bronchial asthma, making the assessment of drug efficacy against COPD difficult
2. Patients using oral corticosteroid medication at a dose in excess of the equivalent 10 mg/day of prednisolon
3. Patients with glaucoma
4. Patients with symptomatic prostatic hypertrophy
5. Patients with hypersensitivity to anticholinergic drugs or powder inhalants
6. Patients with serious complication who are judged by the investigator to be inappropriate as the subjects of study
7. Patients demonstrating clinically problematic abnormal laboratory test values (general blood test, biochemical test, urinalysis). Those showing Glutamic Oxaloacetic Transaminase (GOT) and Glutamic PyruvicTransaminase (GPT) twice the upper limit of the normal range, bilirubin 1.25 times or creatinine 1.25 times of the upper limit of normal range are excluded.
8. Patients with a recent history of myocardial infarction or heart failure (i.e. within 3 months before the screening test)
9. Patients with arrhythmia requiring the treatment with drugs
10. Patients for whom the concomitant use of beta-blocker cannot be prohibited.
11. Patients who began treatment with an ACE inhibitor within 1 month before the screening test
12. Patients with tuberculosis (currently active) or with definite sequela of tuberculosis
13. Patients with a recent history of carcinoma (excluding basal cell carcinoma) (i.e. within the past 5 years)
14. Patients with a history of cystic fibrosis and bronchiectasis
15. Patients with recent onset of upper airway infection (i.e. within 1 month before the screening test)
16. Patients who have taken an investigational drug within one month or within period six times of half-lives of that drug (whichever is longer) before the screening test.
17. Women who are pregnant or who may become pregnant, or those breast feeding
18. Other than above, those who are judged by the investigator to be inappropriate as the subjects of study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2000-09; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events | up to 52 weeks
Changes from baseline in Blood Pressure / Heart Rate | up to 52 weeks
Changes from baseline in ECG | up to 52 weeks
Changes from baseline in laboratory tests | up to 52 weeks

SECONDARY OUTCOMES:
Changes from baseline in Trough Forced expiratory volume in one second (FEV1.0) response | week 24 and 52
Changes from baseline in FEV1.0 at 1 hr post-dosing | week 24 and 52
Changes from baseline in Trough Forced vital capacity (FVC) response | week 24 and 52
Changes from baseline in FVC at 1 hr post-dosing | week 24 and 52
Changes from baseline COPD clinical symptoms (Cough frequency, sputum amount, severity of short breath, nocturnal sleep) | up to 52 weeks
Frequency of rescue use of β2 stimulants | up to 2 weeks
Changes from baseline in Quality of Life QOL (St George's Respiratory Questionnaire (SGRQ) and Airways Questionnaire-20 (AQ20), if possible) | week 24 and 52
Patient's impression | week 24 and 52
Physician's global evaluation | week 24 and 52